CLINICAL TRIAL: NCT00875368
Title: Maraviroc Immune Recovery Study, A Multicenter, Randomized, Placebo-controlled, Exploratory Mechanistic Study Into the Role of Maraviroc on Immune Recovery
Brief Title: Maraviroc Immune Recovery Study
Acronym: MIRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: S.F.L. van Lelyveld (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); Onze Lieve Vrouwe Gasthuis (Other); Slotervaart Hospital (Other); Rijnstate Hospital (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, S.F.L. van Lelyveld, Coordinating investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-283
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: HIV-1; HAART; CD4 cell; Immunologic non-responders; Immunology; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Active Comparator)
  Interventions: Drug: maraviroc
- Placebo (Placebo Comparator): Placebo drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: maraviroc — maraviroc dose dependent on co-medication
  Other Names: Celsentri; Celsentry
  Arms: Maraviroc
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
Rationale: Improving cellular immunity by means of increasing CD4 cells is one of the goals of antiretroviral therapy in HIV, which is achieved by means of virological suppression. A certain group of patients, the so called "immunologic non responders", fail to reach an acceptable CD4 cell increase despite an adequate virologic response on antiretroviral treatment. Recently a new antiretroviral agent, maraviroc (Celsentry®), is registered for the treatment of patients infected with CCR5 tropic HIV-1 virus. However, data is available suggesting that treatment with maraviroc leads to immune recovery (increase in CD4 cells) in patients who are infected with dual/mixed tropic HIV-1 virus, in the absence of a virologic response. This suggests an alternative mechanism for immune recovery, which could be especially beneficial for this group of patients.

Hypothesis: Maraviroc, by a yet unknown mechanism, stimulates immune recovery by increasing CD4+ cell count.

Objective: The primary objective is to confirm the hypothesis that maraviroc stimulates immune recovery; the secondary objective is to explore, by virologic and immunologic investigations, the underlying mechanisms of this hypothesis.

Study design: multicentre, randomized, placebo-controlled, double blind, exploratory mechanistic study.

Study population: HIV-1 infected patients 18 years or older, who meet the inclusion criteria.

Intervention: One group receives maraviroc (dose dependent on co-medication), the other group placebo.

Main study parameters/endpoints: A 30% increase in CD4 cell rise in the treatment group (compared with placebo).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

1. In the treatment group subjects will start with a registered antiretroviral agent (maraviroc).
2. During the treatment year patients will perform several study visits, probably three more compared with regular visits on the outpatient clinic.
3. Each visit, blood will be drawn by venepuncture for immunologic and virologic investigations (see flow chart).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* HAART with a maximal treatment interruption of two weeks
* viral suppression (< 50 copies/ml) for 6 months
* And either:

  * CD4+ count < 200 cells/microliter after minimal one year of treatment with HAART (study group one) OR
  * a CD4+ cell count between 200 and 350 cells/microliter after minimal two years of treatment with HAART (study group two)

Exclusion Criteria:

* HAART consisting of a combination of tenofovir and didanosine
* Active infection for which antimicrobial treatment
* Acute hepatitis B or C
* Chronic hepatitis B or C for which treatment with (peg)interferon and/or ribavirin (Note: patients with untreated chronic hepatitis B or C can be included)
* Immunosuppressive medication
* Radiotherapy or chemotherapy in the past 2 years
* Pregnancy or breastfeeding an infant
* Subjects with known hypersensitivity to maraviroc or to peanuts, or any of its excipients or dyes as follows:

  * Excipients from tablet: microcrystalline cellulose, dibasic calcium phosphate (anhydrous), sodium starch glycolate, magnesium stearate.
  * Film-coat: [Opadry II Blue (85G20583) contains FD&C blue #2 aluminium lake, soya lecithin, polyethylene glycol (macrogol 3350), polyvinyl alcohol, talc and titanium dioxide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
30% increase in CD4+ cell count after 48 weeks | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andy IM Hoepelman, MD, PhD, Principal Investigator — UMC Utrecht
Locations (10):
- Netherlands (10):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Slotervaartziekenhuis, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Kennemer Gasthuis, Haarlem
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Erasmus MC, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Sint Elisabeth Ziekenhuis, Tilburg
  - Ùniversity Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] van Lelyveld SF, Drylewicz J, Krikke M, Veel EM, Otto SA, Richter C, Soetekouw R, Prins JM, Brinkman K, Mulder JW, Kroon F, Middel A, Symons J, Wensing AM, Nijhuis M, Borghans JA, Tesselaar K, Hoepelman AI; MIRS study group. Maraviroc Intensification of cART in Patients with Suboptimal Immunological Recovery: A 48-Week, Placebo-Controlled Randomized Trial. PLoS One. 2015 Jul 24;10(7):e0132430. doi: 10.1371/journal.pone.0132430. eCollection 2015. PMID 26208341